CLINICAL TRIAL: NCT04433559
Title: Randomized, Double-blind, Two-arms Study With Parallel Groups to Determine the Effect of a Phosphodiesterase Inhibitor for 14 Weeks of Treatment Versus Placebo in Women With FSIAD.
Brief Title: Study of Pharmacological Treatment in Women With Female Sexual Interest/Arousal Disorder (FSIAD).
Acronym: FSIAD
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Lidia Larrañaga (Industry)
Responsible Party: Sponsor-Investigator, Lidia Larrañaga, Clinical Trial Coordinator, Laboratorios LITAPHAR, S.L.
Organization: Laboratorios LITAPHAR, S.L. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LITA-004
Record Dates: First submitted 2020-05-06; First posted 2020-06-16 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Sexual Dysfunctions, Psychological
MeSH Terms: conditions — Sexual Dysfunctions, Psychological | interventions — Tadalafil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group Active Tadalafile (Active Comparator): One oral tablet of 1.5 mg IPDE daily for 14 weeks of treatment.
  Interventions: Drug: Tadalafil 1,5 mg oral tablets
- Group Placebo (Placebo Comparator): One oral tablet of placebo daily for 14 weeks of treatment.
  Interventions: Drug: Placebo oral tablets

INTERVENTIONS:
Drug: Tadalafil 1,5 mg oral tablets — Use of tadalafil in the treatment of FSIAD
  Other Names: Tadalafil
  Arms: Group Active Tadalafile
Drug: Placebo oral tablets — Use of placebo in control group
  Other Names: Placebo
  Arms: Group Placebo

SUMMARY:
This clinical trial is a prospective, randomized, double-blind Phase III study with two arms to determine the efficacy and safety of the use of an IPDE in women with FSIAD.

Patients who meet all inclusion criteria and do not meet any of the exclusion criteria will enter the study and receive active product or placebo for 14 weeks.

Patients will be assigned to each treatment group in a randomized and parallel manner. In addition, all volunteers participating in the study will receive medical advice during the study.

The study will have a duration of minimum of 18 weeks and will consist of 3 periods.

DETAILED DESCRIPTION:
This clinical trial is a prospective, randomized, double-blind Phase III study with two arms to determine the efficacy and safety of the use of an IPDE in women with FSIAD.

Patients who meet all inclusion criteria and do not meet any of the exclusion criteria will enter the study and receive active product or placebo for 14 weeks.

Patients will be assigned to each treatment group in a randomized and parallel manner. In addition, all volunteers participating in the study will receive medical advice during the study.

The study will have a duration of minimum of 18 weeks and will consist of 3 periods

ELIGIBILITY:
Inclusion Criteria:

1. Women between 18 and 65 years old. Women of childbearing age (premenopausal, not surgically sterilized at least 3 months before the Selection Visit) must be used during the study a highly effective contraceptive method such as:

   * contraceptive methods or partner vasectomy, and confirm who are not pregnant by pregnancy test negative in the Selection Consultation.

     2. Signature of the informed consent obtained in writing,including a data protection declaration before the participation in the study.

     3. Women with disorders of interest and sexual arousal diagnosed using a semi-structured questionnaire of 5 questions based on DSM-V criteria.

Exclusion Criteria :

1. The following groups of patients with cardiovascular risk:

   * Patients who had suffered myocardial infarction in the 90s previous days,
   * Patients with unstable angina or angina produced during sexual activity,
   * Patients with heart failure corresponding to class II or higher than the New York Heart Association classification (NYHA) in the previous 6 months,
   * Patients with uncontrolled arrhythmias,
   * Patients who had suffered a stroke in the previous 6 months.
2. Patients with disorders of female sexual arousal of origin neurogenic.
3. Patients with female sexual dysfunction associated with disorders psychiatric.
4. Patients with a partner who suffers from sexual dysfunction.
5. Patients with dysphoric excitation disorder and / or with sensation unpleasant genital thickening.
6. Patients with a history of severe thromboembolic disease, hepatic, renal, or neoplastic.
7. Uncontrolled diabetic patients (HbA1c> 8% in the last control).
8. Patients with depression and / or taking antidepressants.
9. Lactation
10. Hypersensitivity to tadalafil and / or drugs and products related (including excipients of the formulation).
11. Patients undergoing treatment with any form of organic nitrate.
12. Patients on treatment with potent CYP3A4 inhibitors (ritonavir, ketoconazole, itraconazole, clarithromycin, erythromycin, and saquinavir) and strong CYP3A4 inducers (carbamazepine, phenytoin, phenobarbital, St. John's wort, rifampin).
13. Patients who have loss of vision in one eye a consequence of anterior ischemic optic neuropathy not arteritic.
14. Patients with any pelvic surgery in the previous 6 months.
15. Known history of drug and / or alcohol abuse in the 6 months prior to the selection consultation.
16. Participation in another study in the 3 months prior to the consultation of selection.
17. Any illness that, in the investigator's judgment, can interfere with compliance with study procedures or study evaluations.
18. Patient with any medical or surgical condition that may interfere with absorption, distribution, metabolism or excretion of the study drug according to the criteria of the researcher.
19. Patients in judicial or police custody.
20. Patients with difficulties in understanding the language in which they gives the information to the subject.
21. Patients who do not agree to the transmission of their anonymous data regarding the documentation and notification functions.
22. Study center, sponsor or CRO staff, their own researcher or relatives of the same.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-08 (Estimated); Primary Completion 2021-08 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Effect of IPDE (Tadalafile) according to FSFI (Female Sexual Function Index) | 14 weeks
  To determine the effect of IPDE at a dose of 1.5 mg versus placebo in women with disorders of interest and sexual arousal using the FSFI (Female Sexual Function Index).
  FSFI contains 19 questions, with each questions with a value minimum of 0 and maximum of 6 points, beeing 0 the worst scenario y 6 the best scenario.

SECONDARY OUTCOMES:
Comparative IPDE Vs placebo according to FSFI | 14 weeks
  To compare the effect of IPDE with respect to placebo in women with disorders of interest and sexual arousal using the FSFI (Female Sexual Function Index).
  FSFI contains 19 questions, with each questions with a value minimum of 0 and maximum of 6 points, beeing 0 the worst scenario y 6 the best scenario.
Comparaive of IPDE Vs placebo according NSSS-Short (New Sexual Satisfaction Scale) | 14 weeks
  To compare the effect of IPDE with respect to placebo in women with disorders of interest and sexual arousal using the questionnaire "The New Sexual Satisfaction Scale" (NSSS-Short).
  NSSS-Short (New Sexual Satisfaction Scale) contains 7 questions, with each questions with a value minimum of 0 and maximum of 100 points, beeing 0 the worst scenario y 100 the best scenario.
Comparative IPDE Vs placebo according to the TSQM (Treatment Satisfaction questionnaire for Medication) | 14 weeks
  To compare the effect of IPDE with respect to placebo in women with disorders of interest and sexual arousal using the "Treatment Satisfaction questionnaire for Medication" (TSQM) version 1.4.
  TSQM (Treatment Satisfaction questionnaire for Medication) contains 14 questions with each questions with a value minimum of 0 and maximum of 80 points, beeing 0 the worst scenario y 80 the best scenario.
Comparative of IPDE Vs placebo according to number of sexual events | 14 weeks
  To compare the effect of IPDE with respect to placebo in women with sexual interest and arousal disorder by measuring the number of sexual events recorded in the weekly diary.
  The diary will be fullfilled by the women according to the number of sexual events.
Comparative of IPDE Vs placebo according to the sexual satisfaction | 14 weeks
  To compare the effect of IPDE with respect to placebo in women with sexual interest and arousal disorder by measuring the sexual satisfaction of sexual intercourse.
  The scale will contain 3 questions, with a visual analog scale. This visual analog scale will contain a scale with different visual easy identificable progesion faces, from very sad face to very happy face, beeging the first sad face, the no satisfaction point, and the last very happy face the very satisfactory sexual event point.
Comparative of IPDE Vs placebo according to ease of arousal | 14 weeks
  To compare the effect of IPDE with respect to placebo in women with disorder of interest and sexual arousal by measuring the ease of arousal during sexual intercourse determined using an analog visual scale.
  The scale will contain 3 questions, with a visual analog scale. This visual analog scale will contain a scale with different visual easy identificable progesion faces, from very sad face to very happy face, beeging the first sad face, the no satisfaction point, and the last very happy face the very satisfactory sexual event point.

IPD SHARING:
Plan to Share IPD: No